CLINICAL TRIAL: NCT00888459
Title: A Pilot Study to Assess the Effectiveness of the Nicotine Lozenge for Smokeless Tobacco Users
Brief Title: A Pilot Study Evaluating Nicotine Lozenges and Self Help
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Oregon Research Institute (Other)
Responsible Party: Jon Ebbert, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-008574; CA121165
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Results first posted 2010-11-04 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Smokeless Tobacco Use
Keywords: tobacco; chew; nrt; nicotine lozenges; self-help
MeSH Terms: interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active (Active Comparator): Self-help counseling material and 4 mg nicotine lozenges
  Interventions: Drug: nicotine replacement therapy
- 2 (Placebo Comparator): self help counseling material and placebo nicotine lozenges
  Interventions: Drug: placebo NRT

INTERVENTIONS:
Drug: nicotine replacement therapy — 4 mg nicotine lozenges, ad lib, for 12 weeks.
  Other Names: Nicotine Lozenges
  Arms: active
Drug: placebo NRT — Placebo nicotine lozenges
  Other Names: placebo
  Arms: 2

SUMMARY:
The investigators are hypothesizing that by offering both self-help materials and mailed nicotine lozenges we will be able to help increase tobacco abstinence rates among ST users, as well as decrease tobacco withdrawal.

DETAILED DESCRIPTION:
Smokeless tobacco (ST) is a known human carcinogen. Long-term ST use is known to increase the risk for oropharyngeal cancer. Most smokeless tobacco users wish to quit. Assisted-self help interventions (i.e., self-help manual, a targeted video, and two support telephone phone calls) have been shown to be superior to manual-only interventions for increasing tobacco abstinence rates. These interventions lend themselves to widespread dissemination, but abstinence rates at 6 months remains low (21%). Providing nicotine replacement therapy (NRT) to ST users receiving assisted self-help interventions could improve upon these ST abstinence rates. If found to be effective, this intervention may increase the ability to disseminate effective interventions to a population of tobacco users for whom few treatment resources currently exist.

ELIGIBILITY:
Inclusion Criteria:

1. male;
2. ≥18 years of age;
3. report ST as their primary tobacco of use;
4. have used ST daily for the past 6 months;
5. indicate that they want to quit;
6. have been provided with, understand, and have signed the informed consent.

Exclusion Criteria:

1. previously enrolled in a study involving the use of the nicotine lozenge;
2. currently using or have completed using (past 30 days) any other behavioral or pharmacologic tobacco treatment program;
3. currently enrolled in another research study;
4. describe having a medical history of: a) unstable angina; b) myocardial infarction within the past 6 months; c) cardiac dysrhythmia other than medication-controlled atrial fibrillation or PSVT; or d) medically-treated or untreated hypertension with BP ≥ 180 systolic OR ≥ 100 diastolic;
5. have phenylketonuria (PKU) [nicotine lozenges contain aspartame which is metabolized to phenylalanine and not processed in individuals with PKU];
6. have another member of their household already participating in this study;
7. have other medical or psychiatric conditions that would exclude the participant;
8. have a score of ≥ 15 on the Patient Health Questionnaire (PHQ-9) on the phone call pre-screen.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon O Ebbert, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Oregon Research Institute, Eugene, Oregon

REFERENCES:
- [Result] Ebbert JO, Severson HH, Croghan IT, Danaher BG, Schroeder DR. A pilot study of mailed nicotine lozenges with assisted self-help for the treatment of smokeless tobacco users. Addict Behav. 2010 May;35(5):522-5. doi: 10.1016/j.addbeh.2009.12.020. Epub 2010 Jan 4. PMID 20060229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first person was pre-screened on 05/20/08 and the last person was randomized on 09/29/08.
Groups:
- Active: 4 mg nicotine lozenges
- Placebo: placebo nicotine lozenges (similar in appearance to the 4 mg lozenge)
Period: Overall Study
Arm/Group | Active | Placebo
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (16.0) | 42.4 (11.7) | 43.0 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Smokeless tobacco [Mean (Standard Deviation); unit: cans/week] | 3.9 (3.1) | 3.7 (2.1) | 3.8 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tobacco Abstinence
Description: self-reported 7-day point prevalence tobacco abstinence at week 12 (end of treatment)
Time Frame: 12 weeks
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 30 | 30
participants | 14 | 11
Statistical Analysis 1: Comparison: Active vs Placebo; Test type: Superiority or Other; p = .432, Chi-squared

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=30) | Placebo (N=30)
Heartburn (Gastrointestinal disorders) | 3 (3) | 0 (0)
Sleep disturbance (Psychiatric disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No